CLINICAL TRIAL: NCT00965081
Title: A Randomized, Double-Blind Comparison of Duloxetine 30 mg QD and Placebo in Adult Patients With Fibromyalgia
Brief Title: A Study for Adult Patients With Fibromyalgia
Acronym: HMGG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12873; F1J-MC-HMGG (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Results first posted 2011-11-03 (Estimated); Last update posted 2011-11-03 (Estimated); Status verified 2011-09

CONDITIONS: Fibromyalgia, Primary; Fibromyalgia, Secondary
MeSH Terms: conditions — Fibromyalgia | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duloxetine (Experimental)
  Interventions: Drug: Duloxetine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine — 30 milligrams (mg) dose daily (QD) by mouth (po) at the same time each day for 12 weeks
  Other Names: Cymbalta; LY248686
  Arms: Duloxetine
Drug: Placebo — QD po at the same time each day for 12 weeks
  Arms: Placebo

SUMMARY:
The main purpose of this study is to determine if 30 milligrams (mg) of duloxetine is effective in the treatment of fibromyalgia compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Meet study criteria for fibromyalgia diagnosis.

Exclusion Criteria:

* Have previously or are currently taking duloxetine.
* Have been diagnosed with certain psychoses, bipolar or schizoaffective disorder
* Have pain symptoms that are difficult to differentiate from fibromyalgia.
* Have seizure disorder, uncontrolled narrow angle glaucoma, or acute liver injury (such as hepatitis) or severe cirrhosis.
* Have had any primary Axis 1 diagnosis other than major depressive disorder or generalized anxiety disorder within the past year.
* Are pregnant or breast-feeding
* Have a current or previous diagnosis of rheumatoid, infectious or inflammatory arthritis or an autoimmune disease
* Have a regional pain syndrome, failed back syndrome or chronic localized pan related to any past surgery
* Have a serious unstable medical illness
* Have a history of substance abuse or dependence within the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2009-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- Mexico (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mérida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morelia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who enter the study with a diagnosis of major depressive disorder (MDD) and who also meet the predefined blinded criteria for worsening of depression during the acute therapy phase will be rescued to daily duloxetine 60 mg for the remainder of the acute therapy phase.
Groups:
- Duloxetine: Duloxetine 30 milligrams (mg) dose daily (QD) by mouth (po) at the same time each day for 12 weeks
  Participants who enter the study with a diagnosis of major depressive disorder (MDD) will be rescued to duloxetine 60 mg QD if they meet the predefined blinded criteria for worsening of depression.
- Placebo: Placebo (inactive capsules identical in appearance to duloxetine capsules) QD po at the same time each day for 12 weeks
  Participants who enter the study with a diagnosis of MDD will be rescued to duloxetine 60 mg QD if they meet the predefined blinded criteria for worsening of depression.
Period: Overall Study
Arm/Group | Duloxetine | Placebo
Started | 155 (2 randomized participants had no post-baseline measures and are not included in outcome measures.) | 153
Completed | 121 (In addition, 16/17 rescue participants completed study on protocol-specified study medication.) | 110
Not Completed | 34 | 43
Not completed — Adverse Event | 14 | 9
Not completed — Lack of Efficacy | 2 | 5
Not completed — Lost to Follow-up | 4 | 5
Not completed — Physician Decision | 2 | 0
Not completed — Protocol Violation | 2 | 5
Not completed — Sponsor Decision | 1 | 0
Not completed — Withdrawal by Subject | 4 | 7
Not completed — Switched to Rescue Arm | 5 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine | Placebo | Total
Number analyzed (Participants) | 155 | 153 | 308
Age Continuous [Mean (Standard Deviation); unit: Years] | 50.89 (11.90) | 50.72 (12.45) | 50.80 (12.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 147 | 293
  Male | 9 | 6 | 15
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 13 | 12 | 25
  Asian | 3 | 0 | 3
  Black or African American | 6 | 5 | 11
  White | 133 | 136 | 269
Region of Enrollment [Number; unit: Participants]
  Argentina | 40 | 38 | 78
  Israel | 14 | 14 | 28
  Mexico | 42 | 42 | 84
  Puerto Rico | 3 | 3 | 6
  United States | 56 | 56 | 112
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/meters squared (kg/m2)] — BMI is an estimate of body fat based on body weight divided by height squared (kg/m^2).
  kilograms/meters squared (kg/m2) | 28.91 (6.00) | 29.49 (6.90) | 29.20 (6.46)
Brief Pain Inventory (BPI) Average Pain Score [Mean (Standard Deviation); unit: Units on a scale] — The BPI-Modified Short Form is a self-reported scale that measures the severity of pain and the interference of pain on function. Severity scores range from 0 (no pain) to 10 (pain as bad as you can imagine). The BPI Average Pain score assesses severity of average pain in the past 24 hours.
  Units on a scale | 6.50 (1.47) | 6.37 (1.67) | 6.44 (1.57)
Brief Pain Inventory (BPI) Mean Interference Score [Mean (Standard Deviation); unit: Units on a scale] — The BPI Mean Interference Score measures mean interference of pain on function in the past 24 hours on 7 items including general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life. Scores range from 0 (does not interfere) to 10 (completely interferes).
  Units on a scale | 5.97 (2.17) | 5.78 (2.28) | 5.88 (2.23)
Fibromyalgia Impact Questionnaire (FIQ) Total Score [Mean (Standard Deviation); unit: Units on a scale] — The FIQ measures participant status, progress, and outcomes over the past week. It consists of 20 items; the first 11 items measure physical functioning. Each item is rated on a 4-point scale. Items 12 and 13 measure number of days participant felt well and number of days participant felt unable to work due to fibromyalgia symptoms. Items 14-20 are numerical, 11-point scales rating work difficulty, pain, fatigue, morning tiredness, stiffness, anxiety, and depression. The total score ranges from 0 to 80. A higher score indicates a more negative impact.
  Units on a scale | 51.11 (12.17) | 50.44 (13.71) | 50.78 (12.94)
Beck Depression Inventory (BDI) Total Score [Mean (Standard Deviation); unit: Units on a scale] — The BDI-II is a 21-item patient-completed questionnaire designed to assess characteristics of depression. Each item is rated on a 4-point scale (0 = not present; 3 = present in the extreme). This questionnaire was used to rate the severity of depressive symptoms and any improvement during the course of the trial. The total score ranges from 0 to 63; the higher the score, the more severe the depressive symptoms.
  Units on a scale | 15.00 (9.64) | 16.84 (11.47) | 15.92 (10.61)
Clinical Global Impression of Severity (CGI-S) for Depression Score [Mean (Standard Deviation); unit: Units on a scale] — The CGI-S for depression scale evaluates the severity of depression at the time of assessment. The score ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). The CGI-S for depression scale was administered by a study physician in the presence of the participant or after having been in the presence of the participant. Number of Participants: Duloxetine = 153, Placebo = 151; scales incorrectly administered were omitted from summary.
  Units on a scale | 2.30 (1.38) | 2.45 (1.45) | 2.38 (1.42)
Patient's Global Impressions of Severity (PGI-S) Score [Mean (Standard Deviation); unit: Units on a scale] — The PGI-S scale is a participant-rated instrument that measures perceived severity of symptoms. It is a 7-point scale where a score of 1 indicates that the patient is "normal, not at all ill," a score of 4 indicates that the patient is "moderately ill," and a score of 7 indicates that the patient is "extremely ill."
  Units on a scale | 3.74 (1.33) | 3.74 (1.47) | 3.74 (1.40)
Beck Anxiety Inventory (BAI) Total Score [Mean (Standard Deviation); unit: Units on a scale] — The BAI is a 21-item patient-completed questionnaire designed to assess characteristics of anxiety. Each item is rated on a 4-point scale (0 = not present; 3 = present in the extreme). This questionnaire was used to rate the severity of anxiety symptoms and any improvement during the course of the trial. The total score ranges from 0 to 63; the higher the score, the more severe the anxiety symptoms. Number of Participants: Duloxetine = 152, Placebo = 153; scales incorrectly administered were omitted from summary.
  Units on a scale | 14.26 (9.35) | 15.04 (10.69) | 14.65 (10.04)
Diagnosis of Major Depressive Disorder (MDD) [Number; unit: Participants] — The Mini International Neuropsychiatric Interview (MINI)was administered to establish if the participant had MDD.
  Participants
    Diagnosis of MDD | 32 | 37 | 69
    No diagnosis of MDD | 123 | 116 | 239
Diagnosis of Generalized Anxiety Disorder (GAD) [Number; unit: Participants] — The MINI was administered to establish if the participant had GAD.
  Participants
    Diagnosis of GAD | 11 | 8 | 19
    No diagnosis of GAD | 144 | 145 | 289

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 12-Week Endpoint in the Brief Pain Inventory (BPI) "24-Hour Average Pain" Item (Question 3) of the BPI-Modified Short Form Score
Description: BPI Average Pain score ranges from 0 (no pain) to 10 (pain as bad as you can imagine). Treatment group difference in Least Squares (LS) Means changes from analysis of covariance (ANCOVA) with terms for treatment group, pooled investigators, baseline. Baseline-observation-carried-forward (BOCF) method used to impute endpoint value for those who discontinued initial double-blind therapy (DBT) due to adverse event (AE); last non-missing observation during initial DBT used to impute missing endpoint for all others. Analyses included all participants having non-missing baseline and endpoint.
Time Frame: Baseline, 12 weeks
Population: Intent-to-treat (ITT) population: all randomized participants. ITT treatment group is group to which participant was randomized regardless of treatment actually received. BOCF method used to impute endpoint value if initial DBT discontinued due to AE. Change from baseline analyses included all those with baseline and ≤1 post-baseline observation.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 153 | 153
Units on a scale | -2.04 (0.20) | -1.70 (0.20)

2. Secondary Outcome: Change From Baseline to 12-Week Endpoint in the Brief Pain Inventory (BPI) - Modified Short Form
Description: BPI-Modified Short Form mean interference score ranges from 0 (does not interfere) to 10 (completely interferes) for pain in past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Treatment group difference in the Least Squares (LS) Means changes from baseline to endpoint is from an analysis of covariance (ANCOVA) with terms for treatment group, pooled investigators and baseline. Last-observation-carried forward (LOCF) endpoint defined as last available post-baseline value obtained during initial double-blind therapy.
Time Frame: Baseline, 12 weeks
Population: Intention to treat (ITT) population: analyses conducted per initial group assignments. The LOCF method was used to impute the missing endpoint during initial double-blind therapy.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 153 | 153
Units on a scale
  Worst Pain | -2.23 (0.23) | -1.98 (0.23)
  Least Pain | -1.56 (0.20) | -1.36 (0.20)
  Pain Right Now | -2.25 (0.23) | -1.90 (0.23)
  Pain Interference - General Activity | -2.19 (0.24) | -1.91 (0.24)
  Pain Interference - Mood | -2.40 (0.24) | -1.82 (0.24)
  Pain Interference - Walking ability | -2.31 (0.22) | -1.74 (0.22)
  Pain Interference - Normal Work | -2.20 (0.24) | -1.77 (0.24)
  Pain Interference - Relations with Other People | -2.05 (0.23) | -1.34 (0.23)
  Pain Interference - Sleep | -2.06 (0.25) | -1.75 (0.25)
  Pain Interference - Enjoyment of Life | -2.48 (0.24) | -1.93 (0.24)
  Mean Interference Score | -2.28 (0.20) | -1.78 (0.20)

3. Secondary Outcome: Patient Global Impression - Improvement (PGI-I) at Endpoint
Description: The PGI-I scale is a patient-rated instrument that measures perceived improvement in symptoms. It is a 7-point scale: score of 1 is "very much better," 4 is "no change," and 7 is "very much worse." Treatment group difference in Least Squares (LS) Means at endpoint is from an analysis of covariance (ANCOVA); model included terms for treatment group, pooled investigators and baseline PGI-Severity (PGI-S).
Time Frame: 12 weeks
Population: Intention to treat (ITT) population: analyses conducted per initial group assignments. The last-observation-carried-forward (LOCF) method was used to impute the missing endpoint during initial double-blind therapy.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 153 | 153
Units on a scale | 2.97 (0.12) | 3.35 (0.12)

4. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I) for Depression at Endpoint
Description: The CGI-I measures clinician's perception of patient improvement at time of assessment compared with start of treatment. Scores range from 1 (very much improved) to 7 (very much worse).
  The treatment group difference in Least Squares (LS) Means at endpoint is from an analysis of covariance (ANCOVA). The model included terms for treatment group, pooled investigators and baseline CGI-Severity (CGI-S).
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 152 | 153
Units on a scale | 3.34 (0.09) | 3.51 (0.09)

5. Secondary Outcome: Change From Baseline to 12-Week Endpoint Beck Depression Inventory-II (BDI-II)
Description: The BDI-II is a 21-item, patient-completed questionnaire to assess characteristics of depression. Each of the 21 items corresponding to a symptom of depression is summed to give a single score. There is a 4-point scale for each item ranging from 0 to 3 (0 = not present; 3 = present in the extreme). The treatment group difference in the Least Squares (LS) Means change from baseline to endpoint is from an analysis of covariance (ANCOVA). The model included terms for treatment group, pooled investigators and baseline.
Time Frame: Baseline, 12 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 140 | 134
Units on a scale | -5.47 (0.60) | -3.91 (0.61)

6. Secondary Outcome: Change From Baseline to 12-Week Endpoint Fibromyalgia Impact Questionnaire (FIQ)
Description: FIQ is a 20-item self-administered questionnaire that measures fibromyalgia (FM) patient status, progress, and outcomes over the past week. The total score ranges from 0 to 80 with higher scores reflecting a more negative impact of FM. The treatment group difference in the Least Squares (LS) Means change from baseline to endpoint is from an analysis of covariance (ANCOVA). The model included terms for treatment group, pooled investigators and baseline.
Time Frame: Baseline, 12 weeks
Population: Intention to treat (ITT) population: analyses conducted per randomly assigned groups. Baseline-observation-carried-forward (BOCF) method used to impute endpoint value for those who discontinued initial double-blind therapy(DB) due to adverse event; last non-missing observation during initial DB used to impute the missing endpoint for all others.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 153 | 153
Units on a scale | -14.62 (1.38) | -9.75 (1.38)

7. Secondary Outcome: Change From Baseline to 12-Week Endpoint Beck Anxiety Inventory (BAI)
Description: The BAI is a 21-item patient-completed questionnaire designed to assess the characteristics of anxiety. Each item is rated on a 4-point scale (0=not present; 3=present in the extreme). The total score ranges from 0 to 63; the higher the score, the more severe the anxiety symptoms.
  The treatment group difference in the Least Squares (LS) Means at endpoint is from an analysis of covariance (ANCOVA). The model included terms for treatment group, pooled investigators and baseline.
Time Frame: Baseline, 12 weeks
Population: Intention to treat (ITT) population: analyses conducted per initial group assignments. The last-observation-carried-forward (LOCF) method used to impute the missing endpoint during initial double-blind therapy.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 138 | 132
Units on a scale | -3.76 (0.67) | -3.31 (0.68)

8. Secondary Outcome: Change From Baseline to 12-Week Endpoint 36-Item Short-Form Health Survey (SF-36)
Description: SF-36 has 36 items with 8 domains: physical functioning, social functioning, bodily pain, vitality, mental health, role-physical, role-emotional, general health; each scored on 0 to 100 scale. Higher scores indicate better status. Mental component summary (MCS) and physical component summary (PCS) based on 8 SF-36 domains. Scales scored using norm-based methods; mean is 50 and standard deviation is 10 in U.S. population. Treatment group difference in Least Squares (LS) Means at endpoint from analysis of covariance. Terms for treatment group, pooled investigators, baseline in model.
Time Frame: Baseline, 12 weeks
Population: Intention to treat (ITT) population: analyses conducted per initial group assignments. The last-observation-carried-forward (LOCF) method used to impute the missing endpoint.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 153 | 153
Units on a scale
  Bodily Pain Transformed (n=141, n=135) | 17.06 (1.87) | 14.01 (1.89)
  General Health Transformed (n=140, n=134) | 7.88 (1.47) | 6.12 (1.50)
  Mental Health Transformed (n=141, n=135) | 9.36 (1.56) | 5.55 (1.59)
  Physical Functioning (n=141, n=135) | 9.53 (1.74) | 6.34 (1.76)
  Role-Emotional (n=141, n=135) | 18.88 (3.45) | 10.69 (3.50)
  Role-Physical (n=141, n=135) | 18.55 (3.48) | 13.13 (3.52)
  Social Functioning (n=141, n=135) | 14.05 (1.93) | 6.75 (1.95)
  Vitality (n=141, n=135) | 11.87 (1.73) | 7.59 (1.74)
  Mental Component (n=140, n=134) | 5.56 (0.85) | 2.87 (0.87)
  Physical Component (n=140, n=134) | 4.75 (0.72) | 3.91 (0.73)

9. Secondary Outcome: Number of Participants With Suicidal Behaviors and Ideations Collected by Columbia -Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is a scale capturing occurrence, severity, and frequency of suicide-related thoughts and behaviors. The number of participants with suicidal behaviors and ideations are provided.
  Suicidal behavior: a "yes" answer to any of 5 suicidal behavior questions which include: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide.
  Suicidal ideation: a "yes" answer to any 1 of 5 suicidal ideation questions which include wish to be dead and 4 different categories of active suicidal ideation.
Time Frame: Baseline through 12 weeks
Population: Only participants having at least 1 post-baseline C-SSRS assessment were included in this analysis.
Measure: Number; unit: Participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 152 | 153
Participants
  Wish to be dead | 3 | 3
  Non-specific active suicidal thoughts | 1 | 0
  Active suicidal ideation with no intent to act | 1 | 0
  Active suicidal ideation, some intent, no plan | 0 | 0
  Active suicidal ideation with specific plan/intent | 0 | 0
  Suicidal behavior - Preparatory acts or behavior | 0 | 0
  Suicidal behavior - Aborted attempt | 0 | 0
  Suicidal behavior - Interrupted attempt | 0 | 0

ADVERSE EVENTS:
Groups:
- Placebo: Placebo (inactive capsules identical in appearance to duloxetine capsules) daily by mouth at the same time each day for 12 weeks.
- Duloxetine 30 mg: Duloxetine 30 mg dose daily by mouth at the same time each day for 12 weeks
- Duloxetine 60 mg: Participants who enter the study with a diagnosis of major depressive disorder (MDD) and who also meet the predefined blinded criteria for worsening of depression during the acute therapy phase will be rescued to daily duloxetine 60 mg for the remainder of the acute therapy phase.
Arm/Group | Placebo | Duloxetine 30 mg | Duloxetine 60 mg
Serious Adverse Events (participants affected / at risk) | 1/153 | 0/155 | 0/17
Other Adverse Events (participants affected / at risk) | 78/153 | 100/155 | 5/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=153) | Duloxetine 30 mg (N=155) | Duloxetine 60 mg (N=17)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=153) | Duloxetine 30 mg (N=155) | Duloxetine 60 mg (N=17)
Palpitations (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 4 (4) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 6 (6) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 5 (5) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (8) | 7 (7) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 13 (13) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (7) | 33 (33) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 3 (3) | 0 (0)
Chills (General disorders) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 4 (4) | 0 (0)
Feeling jittery (General disorders) | 1 (1) | 3 (3) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 3 (4) | 0 (0)
Nasopharyngitis (Infections and infestations) | 7 (7) | 4 (4) | 0 (0)
Pharyngitis (Infections and infestations) | 5 (5) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 3 (3) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (5) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 7 (7) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 6 (6) | 11 (12) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 15 (17) | 21 (21) | 1 (1)
Migraine (Nervous system disorders) | 2 (3) | 3 (3) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 4 (4) | 0 (0)
Sedation (Nervous system disorders) | 1 (2) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 4 (4) | 9 (9) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (4) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 8 (8) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less